CLINICAL TRIAL: NCT07238153
Title: Promoting Emotional and Autonomic Control Through Guided Breathing Exercises for Emerging Adults With Autism
Acronym: PEACE-A
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S70725
Record Dates: First submitted 2025-09-19; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-07

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: Heart rate variability; Stress; Biofeedback; Autism; Movement behavior; Guided breathing exercise; slow paced breathing
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The study begins with an assessment at T0, followed by a five-week baseline period. The assessment consist of a physiological measurement and three mental health questionnaires. During the baseline period, all participants will wear an accelerometer to monitor their movement behaviors. The accelerometer will be wrist worn for 7 consecutive days. After this baseline period, participants will be randomly assigned to one of two intervention groups (HRV- biofeedback or slow-paced breathing) and the second assessment will take place at T1. The following intervention period lasts five weeks. During this period, all participants will receive 3 supervised sessions with the researcher, combined with home-based practice.
  After the intervention period the third assessment will take place at T2. Following the intervention, there will be a five-week no-intervention period for all participants. After this, a follow-up assessment will take place at T3.
Masking Description: The researcher plays an active role during the intervention, and participants will be informed about the different interventions provided in both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slow paced breathing (SPB) (Active Comparator): The participants will receive a 5-week training, starting with one visit to explain the procedure and determine the individual resonance frequency (for reasons of comparison). Afterwards, participants are instructed to practice at home, using the Pebbles. The breathing frequency of the Pebbles will be set at 6 breaths/minute (3-1-4-2) (slow-paced breathing) and participants are instructed to practice 4x5 minutes a day. In week 2 and week 3, follow-up sessions will be scheduled with each participant (in line with the protocol for the HRV-BF group). Similar to the HRV-BF group, the participants will be asked to rate the level of comfort during the training via a secure web-based application (m-path, KU Leuven) and compliance and physiological data will be captured with the Pebbles. The device used to support the home-based training.
  Interventions: Device: Guided breathing exercise - SPB
- Heart rate variability biofeedback (HRV-BF) (Active Comparator): The participants will follow a fixed scheme: consisting of 3 supervised sessions (30 minutes) combined with home-practice on the other days (20 minutes, 4x5 minutes/day), followed by a training period of 2 weeks, without supervised sessions. In the first session, the personal resonance frequency of the participant will be determined. The resonance frequency refers to a breathing frequency between 4.5 and 7 breaths per minute at which heart rate and the breathing pattern are in phase, also known as Respiratory Sinus Arrhythmia. This introductory session is followed by two supervised training session in week 2 and 3. The participants will be asked to rate the level of comfort during the training via a secure web-based application (m-path, KU Leuven) and compliance and physiological data will be captured with the Pebbles. The device used to support the home-based training.
  Interventions: Device: Guided breathing exercise - HRV-BF

INTERVENTIONS:
Device: Guided breathing exercise - SPB — Guided breathing exercises are performed at a fixed pace of 6 breaths per minute (SPB) .
  Arms: Slow paced breathing (SPB)
Device: Guided breathing exercise - HRV-BF — Guided breathing exercises are performed at each participant's individually determined resonance frequency, which typically falls between 4.5 and 7 breaths per minute (HRV-BF).
  Arms: Heart rate variability biofeedback (HRV-BF)

SUMMARY:
This study examines the impact of guided breathing exercises on stress and heart rate variability (HRV) in autistic young adults. It explores how daily movement behavior (sleep, physical activity and sedentary behavior) influences HRV and to what extent two guided breathing exercises can affect HRV. Additionally, the study investigates how participants perceive the exercises in terms of usability and usefulness.

DETAILED DESCRIPTION:
For many autistic individuals, transitioning into adulthood can be challenging and stressful. This stress often affects their mental health. The autistic community has highlighted the need for better mental health support, including accessible and effective ways to manage stress. Among the non-pharmacological interventions aimed at improving mental health via stress reduction, guided breathing interventions are promising, also on a psychophysiological level. During a stressful situation, internal regulatory processes take place to maintain balance, starting by activating the autonomic nervous system (ANS). Prior work indicates that a dysfunction of the ANS contributes to the heightened mental health challenges observed in autistic individuals. Heart rate variability (HRV), the variation in time between heartbeats, is an physiological index of the functioning of the ANS. The Neurovisceral Integration Theory highlights the role of parasympathetic regulation of the heart rate, associating higher vagally mediated HRV with better health, emotional regulation and executive functioning.In autistic individuals, the overall levels of cardiac vagal modulation are lower compared to neurotypical peers.

To date, research investigating the potential of interventions aimed at increasing HRV in autistic individuals is scarce. Moreover, HRV is influenced by several aspects (e.g., sleep, physical activity) and knowledge on their combined impact is necessary to understand how HRV can be used in research and clinical practice. Therefore, in this project, the investigators will explore the role of physical activity, sedentary behavior, and sleep on HRV and determine what constitutes a significant change in HRV.

The investigators will also examine the psychophysiological effects, feasibility, and acceptability of the two leading protocols in guided breathing interventions (heart rate variability biofeedback and slow-paced breathing). HRV-BF optimizes HRV by guiding individuals to breathe at their resonance frequency, synchronizing heart rate and breathing. SPB prescribes to breathe at a fixed pace of 6 breaths per minute.

ELIGIBILITY:
Inclusion Criteria:

* For participants ≥18 years a voluntary written informed consent and for participants < 18 years a written informed consent from the parents or their legally authorized representative and an informed assent of the participant has been obtained prior to any screening procedures
* Male or Female (biological)
* Between 16 and 25 years old
* Diagnosis of autism as described in the DSM-IV/DSM-5(-TR)

Exclusion Criteria:

* Participant has a history of congenital heart diseases, diagnosed cardiovascular abnormalities or somatic diseases conditions that may interfere with the main outcome measure HRV or with the safe practice of breathing exercises (e.g., uncontrolled epilepsy, severe respiratory illness)
* Presence of contra-indications for participating (intervention and/or assessment): acute agitation and/or severe psychiatric symptoms (psychosis, mania or major depression) and/or active substance use.
* The presence of an intellectual disability, defined as an intelligence quotient < 70, as described in the DSM-IV/DSM-V.
* Insufficient knowledge of Dutch language in order to follow instructions and fill out questionnaires.
* Female who is pregnant.
* Participation in another interventional study, with or without an investigational medicinal product (IMP) or device (IMD).
* The use of medication known to affect cardiac modulation (excluding hormonal contraceptives).
* Hearing- or vision impairment that cannot be corrected to normal functioning.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in cardiac vagal modulation of heart rate based on resting-state HRV. | At all assessment points: at the start of the study (week 0, time point 0) before the intervention (week 5, time point 1) + after 5 weeks of intervention (week 10, time point 2) + after 5 weeks at the follow-up (week 15, time point 3)
  Calculated as (1) a time domain measure (RMSSD: Root Mean Square of Successive Differences). Three-lead electrocardiographic data will be captured using the NeXus-10 MKII biofeedback device and Biotrace+ Software (MindMedia B.V., The Netherlands). Disposable, self-adhesive and pre-gelled electrodes (Kendall™ ECG Electrodes Arbo™ H124SG, Covidien, Ireland) will be used without specific skin preparations at a sampling rate of 256 SPS. For the recording of the breathing frequency, an elastic band with stretch-sensitive sensors and a sampling rate of 32 SPS is placed around the waist.
Change in cardiac vagal modulation of heart rate based on resting-state HRV | At all assessment points: at the start of the study (week 0, time point 0) before the intervention (week 5, time point 1) + after 5 weeks of intervention (week 10, time point 2) + after 5 weeks at the follow-up (week 15, time point 3)
  Calculated as (2) a frequency domain measures (HF-HRV). Three-lead electrocardiographic data will be captured using the NeXus-10 MKII biofeedback device and Biotrace+ Software (MindMedia B.V., The Netherlands). Disposable, self-adhesive and pre-gelled electrodes (Kendall™ ECG Electrodes Arbo™ H124SG, Covidien, Ireland) will be used without specific skin preparations at a sampling rate of 256 SPS. For the recording of the breathing frequency, an elastic band with stretch-sensitive sensors and a sampling rate of 32 SPS is placed around the waist.

SECONDARY OUTCOMES:
Change in mental health indicators | At all assessment points: at the start of the study (week 0, time point 0) before the intervention (week 5, time point 1) + after 5 weeks of intervention (week 10, time point 2) + after 5 weeks at the follow-up (week 15, time point 3)
  (1) Symptom Checklist-90 Revised (SCL-90-R): The Dutch version measures eight dimensions: anxiety (ANG), agoraphobia (AGO), depression (DEP), somatization (SOM), cognitive-performance deficits (IN), interpersonal sensitivity and mistrust (SEN), hostility (HOS), and sleep difficulties (SLA). Each item is rated on a 5-point Likert scale from 1 ("not at all") to 5 ("extremely"). The total score ranges from 90 to 450. The total score provides a general measure of psychological distress. Higher scores indicate more symptoms and distress.
  The scores on the eight dimensions range for ANG between 10 and 50, for AGO between 7 and 35, for DEP between 16 and 80, for SOM between 12 and 60, for IN between 9 and 45, for SEN between 18 and 90, for HOS between 6 and 30 and for SLA between 3 and 15. Higher scores indicate more symptoms and distress.
Change in mental health indicators | At all assessment points: at the start of the study (week 0, time point 0) before the intervention (week 5, time point 1) + after 5 weeks of intervention (week 10, time point 2) + after 5 weeks at the follow-up (week 15, time point 3)
  (2) Depression Anxiety Stress Scales (DASS-21): The Dutch version of the DASS-21 measures the presence of symptoms of depression, anxiety, and stress. In consists of 21 items and takes about 10 minutes to complete. Each item is rated on a 4-point Likert scale from 0 ("did not apply to me at all") to 3 ("applied to me very much, or most of the time"). The scale yields three subscale scores: Depression, Anxiety, and Stress, each based on 7 items. Subscale scores therefore range from 0 to 21. To calculate the scores, the subscale scores are multiplied by two, resulting in a final range of 0 to 42 per subscale. Higher scores indicate greater symptom severity.
Change in mental health indicators | At all assessment points: at the start of the study (week 0, time point 0) before the intervention (week 5, time point 1) + after 5 weeks of intervention (week 10, time point 2) + after 5 weeks at the follow-up (week 15, time point 3)
  (3) Perceived stress scale (PSS-10): The Dutch version of the PSS measures the degree to which situations in one's life are appraised as stressful, that is, how unpredictable, uncontrollable, and overloaded respondents experience their lives. It consists of 10 items and takes maximum 5 minutes to complete. Each item is rated on a 5-point Likert scale ranging from 0 ("never") to 4 ("very often"). Four items are positively stated and are reverse-scored (item 4,5,7 en 8). Total scores range from 0 to 40, with higher scores indicating higher levels of perceived stress
feasibility and acceptability of the HRV-BF and SPB interventions. | For 5 weeks 4 times per day (before and after each sessions) during the intervention phase (between week 5 and week 10)
  The investigators will explore how participants experience the guided breathing protocols, including their usability. This aspect will be assessed through a self-report questionnaire, including the registration of perceived stress before and after each sessions, using a Visual Analogue Scale (VAS) ranging from "none" to "a lot".
feasibility and acceptability of the HRV-BF and SPB interventions. | For 5 weeks 4 times per day during the intervention phase (between week 5 and week 10)
  The investigators will explore how participants experience the guided breathing protocols, including their acceptability. This aspect will be assessed through a self-report questionnaire, including the registration of the overall experience of each session, using a Visual Analogue Scale (VAS) after each session going form "very unpleasant" to "very pleasant".
feasibility and acceptability of the HRV-BF and SPB interventions. | During the intervention phase (between week 5 and week 10) and during the once per week guided intervention sessions at week 5, 6 and 7.
  The investigators will explore how participants experience the guided breathing protocols, including their, safety. This aspect will be assessed though self-report questionnaires, including the registration of adverse events and mild negative reactions.
feasibility and acceptability of the HRV-BF and SPB interventions. | During the guided intervention sessions at week 5, 6 and 7.
  The investigators will explore how participants experience the guided breathing protocols, including their, safety. This aspect will be assessed though through observations and contact with the investigator during the guided intervention sessions
feasibility and acceptability of the HRV-BF and SPB interventions. | During the intervention phase (between week 5 and week 10) and during the once per week guided intervention sessions at week 5, 6 and 7.
  The investigators will explore how participants experience the guided breathing protocols, including their, safety. This aspect will be assessed though the registration of adverse events and mild negative reactions.
feasibility and acceptability of the HRV-BF and SPB interventions. | At time point 3 (week 15) during the follow-up assessment
  The investigators will explore how participants experience the guided breathing protocols, including their acceptability, safety, usability and adaptability to daily life. These aspects will be assessed through in-depth interviews. The interview guide was developed based on the Theoretical Framework of Acceptability (TFA). This framework allows for a comprehensive exploration of intervention acceptability through seven key constructs (affective attitude, burden, ethicality, intervention coherence, opportunity costs, perceived effectiveness, and self-efficacy).
Feasibility and acceptability of the HRV-BF and SPB interventions. | At time point 3 (week 15) during the follow-up assessment
  The investigators will explore how participants experience the guided breathing protocols, including their usability. This aspect will be assessed through a self-report questionnaire, namely: the System Usability Scale (SUS), which will provide insight into the usability of the digitally delivered home-based training. Each item will be scored on a five-point Likert scale ranging from "strongly disagree" to "strongly agree. The item scores are summed to calculate the total SUS score, which ranges from 0 to 100, representing the overall system usability. Overall scores from 0 to 50 indicate "not acceptable," 51 to 70 indicate marginal level of usability, and 71 to 100 indicate "acceptable" levels of usability.

CONTACTS AND LOCATIONS:
Overall Officials: Tine Van Damme, Prof. dr., Principal Investigator — KU Leuven
Locations (2):
- Belgium (2):
  - KU Leuven, Leuven, Vlaams Brabant
  - UPC Z.Org, Leuven

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (demographics, primary and secondary outcome measures, adverse events) will be shared. No directly identifying information will be included. The interview questions will be shared, but interview responses will not be made available in order to protect participant privacy.
  The study protocol, the statistical analysis plan, analytic code, and a blank informed consent form will be shared. The de-identified dataset will be accompanied by clear documentation explaining the variables, coding, and outcome measures so that researchers can interpret the data without access to the full protocol or analysis plan.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD will be made available beginning 6 months after publication of the primary results and will remain available for at least 10 years.
Access Criteria: De-identified individual participant data will be shared with qualified researchers for non-commercial scientific purposes. Requests must include a short proposal describing the planned analyses. Access will be granted following review by the principal investigator. Approved researchers will be required to sign a data use agreement prior to receiving access through the KU Leuven Research Data Repository.